CLINICAL TRIAL: NCT06554210
Title: Epidemiological Study of the Markers of Aging in the Cohort of Patient HIV in Brest
Acronym: VIHVA
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: VIHVA 2016.CE31
Record Dates: First submitted 2018-10-01; First posted 2024-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Aging, Premature; HIV Infections
Keywords: Aging; HIV
MeSH Terms: conditions — Aging, Premature; HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
RATIONALE: HIV pathology has been associated with accelerated aging of the infected organism, with no known knowledge of virus, immunosuppression, immune response stimulation, antiretroviral toxicity, and "classic" risks. The data are in good standing from a multicenter cohort with high statistical power but very heterogeneous and not exhaustive. A complementary approach by small, comprehensive cohorts is desirable.

POPULATION CONCERNED: HIV-positive persons OBJECTIVE To describe the aging of the physiological functions of people living with HIV.

SECONDARY OBJECTIVES Assess the determinants (virus / HAART / Immunity / environment) Compare to the general population (historical comparisons) Compare to main body functions MAIN EVALUATION CRITERIA respiratory functional tests, memory test, IMTc, ECG, creatininemia, cancer, Fibroscan, bone densitometry...

SECONDARY EVALUATION CRITERIA Age, sex, phototype, CD4 lymphocytes count, viral load, nadir CD4, antiretroviral exposure, alcohol, tobacco ...

METHODOLOGY Monocentric retrospective study STATISTICS Frailty model, chi2 test, test U INCLUSION CRITERIA Seropositive for HIV, age>18 years Follow-up at least once in the Internal Medicine department between 1995 and 2018 CRITERIA OF EXCLUSION Refusal of the patient or unreachable patient NUMBER OF PATIENTS Between 200 and 300 CALENDAR Duration of inclusions: 3 months Duration of participation of the patient: 20 years (retrospectives ...) Duration of the study: 1 year

DETAILED DESCRIPTION:
Rational:

HIV pathology has been associated with an accelerated aging of the infected organism, without anyone knowing how to do it:

* the direct toxicity of the virus;
* CD4 immuno-depletion and its corollary of opportunistic infections, modification of microbiota, ... ;
* Reactive immune stimulation with chronic inflammation;
* the toxicity of antiretrovirals, particularly nucleoside analogues, responsible for acquired mitochondrial cytopathy;
* And, finally, specific environmental factors related to either the mode of acquisition of the infection (transfusion, drug addiction ...), or the frailty induced by the pathology (psychic or social).

The discordant data of the great cohorts must be supported by cohorts of smaller sizes, more exhaustive, both in item and data, more homogeneous in their social determinants.

Population and Methods:

This retrospective monocentric epidemiological study has several objectives:

* Description of the aging of the population followed on several organs
* Comparison with the data of the closest general population geographically, sociologically and temporally;
* Comparison of the relative age of the different organs with each other: synchronous aging or not?
* Evaluation of a screening / surveillance strategy adapted to local epidemiology

  1. Collect aging data from the functions:

     Kidney: creatinine, calculated clearance of creatinine, microalbuminuria Liver: cytolysis, cholestasis, Fibroscan * pulmonary: pulmonary function tests Heart: ultrasound, ECG Brain: memory disorder screening test Psychism: depression test Musculoskeletal: Bone Densitometry, Calcium, Phosphoremia, Vitamin D Vascular: carotid intima-media thickness
  2. Evaluate the potential determinants:

     Demographic: gender, age, phototype Viral: subtypes, time to infection, undetectable delay, viral load zenith Immune: lymphocyte immunophenotyping, nadir CD4 Iatrogen: antiretrovirals (year / patient exposure, compliance), other treatment Toxic: self-administered questionnaire (alcohol, tobacco and others), expired Hb CO, gammaGT, urinary toxicity test
  3. Correlate aging data of each organ with determinants, correlate between organs with and without adjustment to determinants
  4. Look for the closest population data in the literature and compared with those of the VIHVA cohort.

Ethical considerations:

The data of VIHVA study, approved by the local ethics committee (CCPPRB), was collected upon obtaining the non-opposition of patients.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive persons followed in Internal Medicine departement of Brest University Hospital

Exclusion Criteria:

* opposition of the study
* <18 ans

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All persons followed between 2003 to 2018 in the one center (Internal Médicine) of the West Brittany cohort
Sampling Method: Non-Probability Sample
Enrollment: 213 (Actual)
Dates: Start 2017-01-08 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
renal aging | yearly
  creatinin level, creatinin clearance, microalbuminuria
pulmonary aging | at last one
  respiratory functional test
liver aging | at last one
  elastometry (Fibroscan*)
neurological aging | at last one
  memory tests
vascular aging | at last one
  intima-media thickness, systolic and diastolic blood pressure
Bone aging | at last one
  osteodensitometry
heart aging | at last one
  ECG, echography

CONTACTS AND LOCATIONS:
Overall Officials: Luc de Saint-Martin, MD, PhD, Study Director — University Hospital, Brest
Locations (1):
- Internal Medicine Department of University Hospital, Brest, France